CLINICAL TRIAL: NCT06217016
Title: Effect of Intermittent Urethral Catheter Clamping Combined With Active Urination Training (ICCAUT) Strategy on Postoperative Re-catheterization Secondary to Urinary Retention After Radical Rectal Cancer Surgery (ICCAUT-2)
Brief Title: Effect of ICCAUT Strategy on Postoperative Urinary Retention After Radical Rectal Cancer Surgery (ICCAUT-2)
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The ICCAUT-1 trial failed to demonstrate the superiority of the ICCAUT strategy in urinary dysfunction. Therefore, there is no need to conduct subsequent trials.
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yuchen Guo, Ph.D., Prof., The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ICCAUT -2
Record Dates: First submitted 2024-01-05; First posted 2024-01-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Urinary Retention; Rectal Cancer; Urinary Catheterization
Keywords: urinary retention; rectal cancer; bladder training
MeSH Terms: conditions — Urinary Retention; Rectal Neoplasms

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Masking Description: The patients and bedside nurses cannot be blinded, but the attending physicians and the medical ultrasound doctor will be blinded. The medical team will ensure that the patients and bedside nurses keep the group assignment confidential from the attending physicians and the medical ultrasound doctor. Unblinding will occur when the patient is discharged, and any instances of premature unblinding will be recorded. Additionally, the data analysts involved in this study will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ICCAUT Group (Experimental): Patients undergoing laparoscopic/robotic rectal cancer TME surgery will undergo bladder training. The bladder training include intermittent catheter clamping and active urination to facilitate complete bladder emptying each time the catheter is released, which we called ICCAUT strategy. The training will commence at 9:00 am on the first postoperative day, and the catheter will be removed at 9:00 am on the second postoperative day.
  Interventions: Procedure: ICCAUT
- Free Drainage Group (Other): Patients undergoing laparoscopic/robotic rectal cancer TME surgery will have their urinary catheter kept open postoperatively, and the catheter will be removed at 9:00 am on the second postoperative day.
  Interventions: Procedure: Free drainage

INTERVENTIONS:
Procedure: ICCAUT — In this study ,the ICCAUT strategy include intermittent catheter clamping and active urination training. For patients in the ICCAUT group, intermittent catheter clamping will be initiated at 9:00 AM. The catheter will be clamped for 3 h, followed by a 5-minute release, which is one cycle. The next cycle will begin after the cycle was completed. Catheter training is to conclude at 10:00 PM on the first postoperative day, and the catheter is left open during the night. At 6:00 AM on the second postoperative day, another cycle of catheter training will be performed, with the catheter removed at 9:00 AM. During the training period, if the patient experiences a strong urge to urinate before the 3-hour clamping time is over, the clamping can be released in advance for 5 min, allowing the patient to proceed to the next cycle of bladder training. Each time the catheter is released, we will encourage the patients to actively initiate urination to facilitate complete bladder emptying.
  Arms: ICCAUT Group
Procedure: Free drainage — For patients in the free draining group, no intervention will be performed on the catheter during this period. The catheter will be removed at 9:00 AM on postoperative day two.
  Arms: Free Drainage Group

SUMMARY:
The objective of this trial is to investigate the effect of bladder training on the incidence of re-catheterization after proctectomy. In this study, the bladder training include intermittent urethral catheter clamping combined with active urination training, which we called ICCAUT strategy. This prospective, single-center, randomized controlled trial will enroll patients with rectal cancer who will be randomized in a 1:1 ratio to the ICCAUT group or the free-drainage group. In the ICCAUT group, patients will undergo intermittent clamping of the urinary catheter before its removal. Each time the catheter is released, we will encourage the patients to actively initiate urination to facilitate complete bladder emptying. While patients in the free-drainage group will not undergo any specific training. The urinary catheter will be removed on the second postoperative day for both groups. The primary endpoint is the incidence of re-catheterization due to urinary retention. Secondary endpoints include urinary tract infection (UTI), time of first urination after catheter removal, residual urine volume after the first urination, postoperative morbidity and mortality within 30 days, as well as urinary function within 30 postoperative days.

DETAILED DESCRIPTION:
Urinary catheter placement is a standard procedure before proctectomy. However, the necessity of bladder training prior to catheter removal remains uncertain. The objective of this trial is to investigate the effect of bladder training on the incidence of re-catheterization after proctectomy. In this study, the bladder training include intermittent urethral catheter clamping combined with active urination training, which we called ICCAUT strategy. This prospective, single-center, randomized controlled trial will enroll patients with rectal cancer who will be randomized in a 1:1 ratio to the ICCAUT group or the free-drainage group. In the ICCAUT group, patients will undergo intermittent clamping of the urinary catheter before its removal. Each time the catheter is released, we will encourage the patients to actively initiate urination to facilitate complete bladder emptying. While patients in the free-drainage group will not undergo any specific training. The urinary catheter will be removed on the second postoperative day for both groups. The primary endpoint is the incidence of re-catheterization due to urinary retention. Secondary endpoints include urinary tract infection (UTI), time of first urination after catheter removal, residual urine volume after the first urination, postoperative morbidity and mortality within 30 days, as well as urinary function within 30 postoperative days.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a confirmed preoperative diagnosis of rectal cancer.
2. Patients with tumors located below the rectosigmoid junction, as determined by preoperative computed tomography (CT) or rectal magnetic resonance imaging (MRI).
3. Patients undergoing laparoscopic or robotic-assisted total mesorectal excision (TME) for rectal cancer.

Exclusion Criteria:

1. History of abdominal surgery involving the rectum, sigmoid colon, left hemicolectomy, bladder resection or partial resection, prostate surgery, or hysterectomy.
2. History of urethral injury, cranial surgery, spinal surgery, stroke with limb dysfunction, or Parkinson's disease.
3. Inability to urinate through the urethra preoperatively due to various reasons (e.g., ureteral puncture or ureterostomy).
4. Presence of urinary tract infection preoperatively.
5. Previously diagnosed with bladder overactivity syndrome, urinary retention or voiding dysfunction, or diabetic bladder disease.
6. Concomitant resection of other pelvic organs was performed during surgery, including the bladder, prostate, uterus, cervix, and vagina, except for simple adnexal resection.
7. Lateral lymph node dissection for rectal cancer.
8. Injury to the ureter, bladder, or urethra during the perioperative period.
9. Preoperative renal dysfunction (serum creatinine level >133 μmol/L).
10. Emergency surgery.
11. Male patients with preoperative benign prostatic hyperplasia receiving medication treatment.
12. Patients with a ureteral stent or ureteral stricture, or bilateral hydronephrosis.
13. Conversion to open surgery.

Withdrawal Criteria:

After randomization, patients will be withdrawn from the trial if the following situations occur:

1. Inability to remove the urinary catheter within 5 days postoperatively due to various reasons (e.g., impaired consciousness, transfer to the intensive care unit (ICU), Sequential Organ Failure Assessment (SOFA) score ≥2, etc.).
2. Secondary catheterization was performed after catheter removal for reasons other than urinary retention (e.g., secondary surgery, shock, rectal bladder leakage, ureteral leakage, or urethral injury).
3. Patient requests to withdraw from the study at any time during the entire study process.
4. Selective α1-adrenergic receptor blocker is used during the first catheterization of the patient due to medical necessity.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
secondary catheterization owing to urinary retention | within 7 days after the first time of urethral catheter removal
  The primary endpoint of this study is the rate of secondary catheterization owing to urinary retention until discharge. Secondary catheterization can be performed by urethral catheter insertion or suprapubic puncture. The decision to perform secondary catheterization is based on the specific criteria determined by the clinician.

SECONDARY OUTCOMES:
Urinary tract infections | within 1 days after the first time of urethral catheter removal
  A urinary tract infection is characterized by an inflammatory response in the urinary tract epithelium resulting from bacterial invasion. To diagnose a urinary tract infection, the following criteria must be met simultaneously: 1) urinalysis indicating a bacterial count above the upper limit of normal and 2) positive urine culture.
The time to first voiding after catheter removal | within 1 days after the first time of urethral catheter removal
  The time to first voiding after catheter removal refers to the duration, measured in hours, from the moment the catheter was removed until the patient spontaneously voids for the first time.
The residual urine volume after the first voiding | within 1 days after the first time of urethral catheter removal
  The residual urine volume after the first voiding is determined by assessing the volume of urine remaining in the bladder immediately after the patient's initial voiding following catheter removal using bladder ultrasonography.
Graded assessment of catheter-related bladder discomfort (CRBD) | within 1 days after the first time of urethral catheter removal
  CRBD is a questionnaire given to the patients, to investigate the severity of the discomfort of patients to the urinary catheter
Voiding function | on the second day after the first time of urethral catheter removal, and at the 30th day after surgery
  Voiding function is evaluated by International Consultation on Incontinence Questionnaire-Short Form (ICIQ-SF) and International Prostate Symptom Score (IPSS).
Postoperative complications | within 30 days after the operation
  Complications that occur within 30 days after the operation will be evaluated and documented according to the Clavien-Dindo classification (19). Complications of grade II or higher were analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Yuchen Guo, Ph.D, Principal Investigator — The First Hospital of Jilin University
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: Yes
If other researchers can provide valid reasons or demonstrate a need for additional collaboration, we may consider to share the data upon their request after we complete ours study.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: after we complete ours study.
Access Criteria: Researchers can provide valid reasons or demonstrate a need for additional collaboration with us